CLINICAL TRIAL: NCT03186950
Title: Stainless Steel Crowns Versus Bulkfill Composite Resin for Restoring Primary Molars After Endodontic Treatment: Randomized Clinical Trial
Brief Title: Stainless Steel Crowns Versus Bulkfill Composite Resin for Restoring Primary Molars After Endodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniela Prócida Raggio, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENDOREST
Record Dates: First submitted 2016-07-13; First posted 2017-06-14 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restoration with Stainless Steel Crowns (Active Comparator): Restoration of the tooth after endodontic treatment using stainless steel crown.
  Interventions: Procedure: Restoration with Stainless Steel Crowns
- Restoration using BulkFill CR (Experimental): Restoration of the tooth after endodontic treatment using bulkfill composite resin
  Interventions: Procedure: Restoration using BulkFill CR

INTERVENTIONS:
Procedure: Restoration with Stainless Steel Crowns — After finishing the endodontic treatment with Guedes-Pinto Paste, the restoration of the teeth will be made using Stainless Steel Crowns.
  Arms: Restoration with Stainless Steel Crowns
Procedure: Restoration using BulkFill CR — After finishing the endodontic treatment with Guedes-Pinto Paste, the restoration of the teeth will be made using BulkFill composite resin
  Arms: Restoration using BulkFill CR

SUMMARY:
The pulp therapy in primary teeth is designed to eliminate the infection and keep the tooth in a functional state until its natural exfoliation. An important step for the success of endodontic therapy is the final restoration, which must seal the tooth, avoiding new contamination. Thus, this study proposes to carry out a randomized clinical trial with longitudinal follow-up of two years, in order to compare the degree of success of endodontic treatment in primary teeth restored with two different techniques: composite resin (Filtek Bulk Fill - 3M ESPE) or stainless steel crowns (3M ESPE). Success will be measured by clinical and radiographic features of primary teeth treated with the different restorations after 1, 6, 12 and 24 months. Among the secondary outcomes that will be assessed are the quality and durability of restorations and the cost benefit of treatments. Patients who seek the university clinics and require endodontic treatment will be invited to participate. The sample unit is the tooth and these will be randomized in groups through a randomization list created and distributed in sequential opaque envelopes. The envelope will be opened only after the end of endodontic treatment, to ensure allocation concealment. The data will be statistically analyzed using the Stata 12.0 (Stata Corporation, College Station, TX, USA). The longevity of the treatments will be evaluated by estimating survival rates using the Kaplan-Meier method. Differences between survival rates according to the type of endodontic proposed treatment will be analyzed using the log-rank test. All other clinical variables will be analized using Cox regression. The significance level for all analyzes will be 5%.

DETAILED DESCRIPTION:
The pulp therapy in primary teeth is designed to eliminate the infection and keep the tooth in a functional state until its natural exfoliation. An important step for the success of endodontic therapy is the final restoration, which must seal the tooth, avoiding new contamination. Thus, this study proposes to carry out a randomized clinical trial with longitudinal follow-up of two years, in order to compare the degree of success of endodontic treatment in primary teeth restored with two different techniques: composite resin (Filtek Bulk Fill - 3M ESPE) or stainless steel crowns (3M ESPE). Success will be measured by clinical and radiographic features of primary teeth treated with the different restorations after 1, 6, 12 and 24 months. Among the secondary outcomes that will be assessed are the quality and durability of restorations and the cost benefit of treatments. Patients who seek the university clinics and require endodontic treatment will be invited to participate. The sample unit is the tooth and these will be randomized in groups through a randomization list created and distributed in sequential opaque envelopes. The envelope will be opened only after the end of endodontic treatment (made with Guedes-Pinto paste), to ensure allocation concealment. The data will be statistically analyzed using the Stata 12.0 (Stata Corporation, College Station, TX, USA). The longevity of the treatments will be evaluated by estimating survival rates using the Kaplan-Meier method. Differences between survival rates according to the type of endodontic proposed treatment will be analyzed using the log-rank test. All other clinical variables will be analized using Cox regression. The significance level for all analyzes will be 5%.

ELIGIBILITY:
Inclusion Criteria:

* Remaining tooth structure and location of the lesion allow rehabilitation
* Do not have internal or external resorption involving more than 1/3 the length of the root
* Do not have bone loss in lateral root or crypt disruption
* With the presence of at least half of the root

Exclusion Criteria:

* patients that do not fit the inclusion criteria
* patients whos parents did not sign the assentiment term
* patients with systemic desease

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Endodontic Treatment survival | 12 months
  The primary outcome will be the success or failure of endodontic treatments evaluated through the tooth permanence in the arcade on clinical and radiographic conditions of normality compared between groups restorations (steel crown or composite).
  The clinical criteria to determine success are: absence of fistula, absence of painful symptoms, absence of pathological mobility and adequate gingival contour. Radiographically, the success criteria are: absence / reduction of rarefaction and absence / bone thinning in the furcation region later, maintenance of periradicular space, root resorption compatible with eruptive phase and absence of pathological resorption
Need for new intervention | 12 months
  It will be assess the need for any type of reintervention, both for the steel crown group and for the composite resin. Thus, our primary outcome will be measured in accordance with the evaluation of restorations, not only by the failure or not endodontic treatment.
  Clinical sucess: no fistulae or abscess Radiographic sucess: Reduction or maintenance of the interradicular lesion; No crypt breakup

SECONDARY OUTCOMES:
Cost-efficacy between the groups | baseline, 1, 6, 12 and 24 months
  The cost effectiveness of the restoration will be evaluated through consultation that will be timed and cost form developed for the study.
Acceptance of the treatments | Baseline
  Evaluate the acceptance of the treatments by the patients and their guardians, using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela P Raggio, Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo - School of Dentistry, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coll JA, Sadrian R. Predicting pulpectomy success and its relationship to exfoliation and succedaneous dentition. Pediatr Dent. 1996 Jan-Feb;18(1):57-63. PMID 8668572
- [Background] Garcia-Godoy F. Evaluation of an iodoform paste in root canal therapy for infected primary teeth. ASDC J Dent Child. 1987 Jan-Feb;54(1):30-4. PMID 3468139
- [Background] Rifkin A. A simple, effective, safe technique for the root canal treatment of abscessed primary teeth. ASDC J Dent Child. 1980 Nov-Dec;47(6):435-41. No abstract available. PMID 6934178
- [Background] Rifkin A. The root canal treatment of abscessed primary teeth--a three to four year follow-up. ASDC J Dent Child. 1982 Nov-Dec;49(6):428-31. No abstract available. PMID 6960030